CLINICAL TRIAL: NCT04922684
Title: Can Mimic Emotional Expression Training Help Improve Emotion Processing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-66
Record Dates: First submitted 2021-05-14; First posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Healthy
Keywords: Mimic facial expression training; Autistic trait; Mirror neuron system; Emotion processing; Emotion recognition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lower austic sub-group (Active Comparator): 16 times of mimicking emotional expressions
  Interventions: Behavioral: Mimic facial expressions
- Higher austic sub-group (Experimental): 16 times of mimicking emotional expressions
  Interventions: Behavioral: Mimic facial expressions

INTERVENTIONS:
Behavioral: Mimic facial expressions — 16 times (4 times a week, last 4 weeks) of mimicking facial expressions.

SUMMARY:
The main aim of the present study is to investigate whether mimicking emotional expressions training via FaceReader software can improve emotional processing and recognition in healthy subjects, especially individuals with hityer autistic traits.

DETAILED DESCRIPTION:
Some mood and trait questionnaires such as Autism Spectrum Quotient, Social Responsiveness Scale,State-Trait Anxiety Inventory,Beck's Depression Inventory etc are asked to complete. 90 healthy male subjects will receive 16 times (4 times a week , 4 weeks) of mimicking emotional expressions training via Facereader. During training, 3 times of fNIRS (t2,t9 and t16) were recorded simultaneously. fMRI scanning, including emotion processing and emotion recognition tasks, 7 minutes resting data, ans DTI data will be collected before and after the training. After fMRI scaning, behavioral ratings (i.e. intensity and valence) and eye-tracking data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders

Exclusion Criteria:

* history of head injury;
* pregnant, menstruating, taking oral contraceptives;
* medical or psychiatric illness.

Ages: 17 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Intensity score of subjects' mimic facial emotions | an average of 4 weeks
  The measurement was monitored and analyzed by FaceReader software before and after the 4-week training session and subjects' facial expressions of mimicking certain emotions will be calculated into intensity, ranging from 0 to 1.
Valence score of subjects' mimic facial emotions | an average of 4 weeks
  The measurement was monitored and analyzed by FaceReader software before and after the 4-week training session and subjects' facial expressions of mimicking certain emotions will be calculated into valence, ranging from -1 to 1.
Arousal score of subjects' mimic facial emotions | an average of 4 weeks
  The measurement was monitored and analyzed by FaceReader software before and after the 4-week training session and subjects' facial expressions of mimicking certain emotions will be calculated into arousal, ranging from 0 to 1.
Task-dependent functional MRI data | an average of 4 weeks
  Neural activities of brain regions, notably mirror neuron system will be collected for analysis when the subjects participate in a face processing and emotion recognition task in a MRI scanner before and after the 4-week training session.

CONTACTS AND LOCATIONS:
Overall Officials: Weihua Zhao, Dr., Study Chair — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China, Chengdu, Sichuan, China